CLINICAL TRIAL: NCT00159029
Title: Haplotype Analysis of Alpha Globin Genes in Israeli Ethnic Groups
Brief Title: Genetics of Alpha Thalassemia in Israeli Ethnic Groups
Status: Completed | Type: Observational
Sponsor: Deborah Rund (Other)
Responsible Party: Sponsor-Investigator, Deborah Rund, Senior Hematologist, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Other Study IDs: 152910-HMO-CTIL
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Alpha Thalassemia
MeSH Terms: conditions — alpha-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA isolated from peripheral blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
Alpha thalassemia causes mild anemia and is found in many ethnic groups. Usually it is found in regions where malaria is endemic. We have found that alpha thalassemia is common in Ashkenazim, whose countries of origin are in temperate climates.

We are analyzing the alpha globin genes of individuals of many ethnic groups and will compare to try to define the origin of thalassemia in these individuals of European extraction.

DETAILED DESCRIPTION:
Alpha thalassemia causes mild anemia and is found in many ethnic groups. Usually it is found in regions where malaria is endemic. We have found that alpha thalassemia is common in Ashkenazim, whose countries of origin are in temperate climates.

We are analyzing the alpha globin polymorphisms to determine the haplotypes of individuals of many ethnic groups and will compare to try to define the origin of thalassemia in these individuals of European extraction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of deletional alpha thalassemia

Exclusion Criteria:

* under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to Hadassah Hospital for anemia with microcytosis who are found to have alpha thalassemia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Rund, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Rund D, Filon D, Jackson N, Asher N, Oron-Karni V, Sacha T, Czekalska S, Oppenheim A. An unexpectedly high frequency of heterozygosity for alpha-thalassemia in Ashkenazi Jews. Blood Cells Mol Dis. 2004 Jul-Aug;33(1):1-3. doi: 10.1016/j.bcmd.2004.04.009. PMID 15223003